CLINICAL TRIAL: NCT04122053
Title: Can Including Genotype Information Increase the Effectiveness of Dietary Interventions? Polymorphism of the CYP1A2 Gene and Caffeine Intake in Healthy Adults
Brief Title: Personalized Nutrition Caffeine Intake in Healthy Adults.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poznan University of Life Sciences (Other)
Responsible Party: Principal Investigator, Agata Chmurzyńska, Professor, Poznan University of Life Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: UKB196/19
Record Dates: First submitted 2019-10-03; First posted 2019-10-10 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: CYP1A2 Polymorphism
Keywords: intake; caffeine; coffee; genotype; personalized nutrition
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: eligible volunteers will be randomly assigned to one of the study groups which receive either dietary advice or dietary advice and genotype information
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): group will receive dietary advice and genotype information
  Interventions: Behavioral: Intervention group with genotype information
- Control group (Active Comparator): group will receive dietary advice
  Interventions: Behavioral: Control group without genotype information

INTERVENTIONS:
Behavioral: Intervention group with genotype information — Results of genotyping will be translated into personalised dietary recommendations. Subjects will be informed about their genotypes from the beginning of the study. The importance of personalised recommendations will be explained.
  Arms: study group
Behavioral: Control group without genotype information — Subjects will receive personalised dietary recommendations, but at the beginning they will not be informed about their genotypes and the meaning of personalisation. Information about their genotype will be given to the participants at the and of study.
  Arms: Control group

SUMMARY:
Personalized nutrition is one of the most up to date trends in human nutrition and gains much interest of general public and scientists as well. Although we have gained some knowledge on gene-trait associations, the real effectiveness and usefulness of genotype-based nutritional recommendations is unknown. Many personalized nutrition companies are on the market today, some of them use personalized nutrition based on genotype analysis. For this reason, scientific basis of this approach should be clarified. Moreover, the effect of using genotype information in dietary interventions aimed at decreasing caffeine intake has never been tested. Our project can thus increase knowledge which can be applied in dietary counseling practice. Although we focus on caffeine intake, the study is designed as a proof of concept.

DETAILED DESCRIPTION:
Considering current knowledge and recognizing the existing gaps we hypothesize that providing genotype information may increase adherence to dietary recommendations.

The main aim of the project is thus testing the effectiveness of a genotype-based personalized dietary intervention targeted at decreasing caffeine intake.

Specific aims of the study include:

* Implementation of the application for mobile devices which will be designed to assess caffeine intake.
* Testing whether providing information on CYP1A2 polymorphism affects effectiveness of the dietary intervention aimed at decreasing caffeine intake.
* Testing whether changes in dietary behavior can persist over time To accomplish the study goals a group of healthy adults will be enrolled. Participants will complete an informed consent procedure. As we aim at decreasing caffeine intake, we plan to first screen for people drinking at least 2 cups of coffee or with total caffeine intake over 200 mg/day. Then genotype screening will be performed and eligible volunteers will be randomly assigned to one of the study groups which receive either dietary advice or dietary advice and genotype information.

ELIGIBILITY:
Inclusion criteria:

* age 18-60
* daily coffee intake at a minimum 2 cups (or equivalent total caffeine intake)

Exclusion criteria:

* injuries,
* chronic diseases (e.g. diabetes, metabolic syndrome, cancer, hyperthyroidism),
* recent dieting,
* pregnancy or breastfeeding,
* no caffeine intake,
* taking chronic pain management pills which contain caffeine.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 94 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-02-17 (Actual); Study Completion 2021-02-17 (Actual)

PRIMARY OUTCOMES:
Caffeine intake level from dietary sources | baseline, 20 week
  caffeine intake (mg/day)
frequency of minor allel | Baseline
  genotyping for CYP1A2 polymorphism (rs762551); assessment of possible genotypes (AA, AC, CC) will be performed with the use of TaqMan probes

SECONDARY OUTCOMES:
body mass(BM) | Baseline, 20 weeks
  Changes in BM (kg) within groups and between groups
Fat Free Mass (FFM) | Baseline, 20 weeks
  FFM changes within (kg) groups and between groups
Fat Mass% (FM%) | Baseline, 20 weeks
  FM% changes within groups and between groups
Total cholesterol (TChol) | Baseline, 20 weeks
  Changes in TChol (mg/dl) within groups and between groups
Blood HDL-cholesterol (HDL-C) | Baseline, 20 weeks
  HDL-C (mg/dl) concentrations change within the group and between the groups
Blood LDL-cholesterol (LDL-C) | Baseline, 20 weeks
  LDL-C (mg/dl) concentrations change within the group and between the groups
Blood triacylglycerol (TAG) | Baseline, 20 weeks
  TAG (mg/dl) concentrations change within the group and between the groups
Blood glucose (GLU) | Baseline, 20 weeks
  GLU (mg/dl) concentrations change within the group and between the groups
Insulin (INS) | Baseline, 20 week
  INS (ulU/ml) concentrations change within the group and between the groups
Dietary intake | Baseline
  macro and micronutrient intake (g,mg,ug)
aspartate aminotransferase (ASPAT) | Baseline, 20 weeks
  ASPAT [U/l] Changes within groups and between groups
Alanine transaminase (ALAT) | Baseline, 20 weeks
  ALAT [U/l] Changes within groups and between groups
waist circumference (WC) | Baseline, 20 weeks
  WC (cm) Changes within groups and between groups
hips circumference (HC) | Baseline, 20 weeks
  HC (cm) changes within groups and between groups

CONTACTS AND LOCATIONS:
Overall Officials: Ewa Bulczak, Msc, Principal Investigator — Poznan University of Life Science
Locations (1):
- Poznan University of Life Sciences, Poznan, Poland

IPD SHARING:
Plan to Share IPD: No